CLINICAL TRIAL: NCT04941261
Title: Phase II Clinical Trial to Evaluate the Safety and Immunogenicity of Recombinant Recombinant Norovirus Bivalent (GI. 1 / GII. 4) Vaccine(Hansenula Polymorpha) in Healthy People Aged Aged From 6 Months to 59 Years
Brief Title: Clinical Trial to Evaluate the Recombinant Norovirus Bivalent (GI. 1 / GII. 4) Vaccine (Hansenula Polymorpha)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Vaccine and Serum Institute, China (Industry)
Collaborators: Lanzhou Institute of Biological Products Co., Ltd (Industry); Beijing Zhong Sheng Heng Yi Pharmaceutical Technology Co., Ltd. (Unknown); Zhengzhou University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CXSL1700011-Ⅱ
Record Dates: First submitted 2021-06-18; First posted 2021-06-28 (Actual); Last update posted 2022-10-28 (Actual); Status verified 2022-05

CONDITIONS: Norovirus Infections; Norwalk Gastroenteritis
MeSH Terms: conditions — Caliciviridae Infections | interventions — Vaccines

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (15):
- 18-59 years old group A (Experimental)
  Interventions: Biological: middle-dose Norovirus Bivalent (GI.1 / GII.4) Vaccine
- 18-59 years old group B (Experimental)
  Interventions: Biological: high-dose Norovirus Bivalent (GI.1 / GII.4) Vaccine
- 18-59 years old group C (Placebo Comparator)
  Interventions: Biological: placebo
- 6-17 years old group A (Experimental)
  Interventions: Biological: middle-dose Norovirus Bivalent (GI.1 / GII.4) Vaccine
- 6-17 years old group B (Experimental)
  Interventions: Biological: high-dose Norovirus Bivalent (GI.1 / GII.4) Vaccine
- 6-17 years old group C (Placebo Comparator)
  Interventions: Biological: placebo
- 3-5 years old group A (Experimental)
  Interventions: Biological: middle-dose Norovirus Bivalent (GI.1 / GII.4) Vaccine
- 3-5 years old group B (Experimental)
  Interventions: Biological: high-dose Norovirus Bivalent (GI.1 / GII.4) Vaccine
- 3-5 years old group C (Placebo Comparator)
  Interventions: Biological: placebo
- 6-35 months old group A (Experimental)
  Interventions: Biological: middle-dose Norovirus Bivalent (GI.1 / GII.4) Vaccine
- 6-35 months old group B (Experimental)
  Interventions: Biological: high-dose Norovirus Bivalent (GI.1 / GII.4) Vaccine
- 6-35 months old group C (Placebo Comparator)
  Interventions: Biological: placebo
- 6-35 months old group D (Experimental)
  Interventions: Biological: middle-dose Norovirus Bivalent (GI.1 / GII.4) Vaccine
- 6-35 months old group E (Experimental)
  Interventions: Biological: high-dose Norovirus Bivalent (GI.1 / GII.4) Vaccine
- 6-35 months old group F (Placebo Comparator)
  Interventions: Biological: placebo

INTERVENTIONS:
Biological: middle-dose Norovirus Bivalent (GI.1 / GII.4) Vaccine — Intramuscular injection of middle-dose Norovirus Bivalent (GI.1 / GII.4) Vaccine in the deltoid muscle of the upper arm
  Arms: 18-59 years old group A; 3-5 years old group A; 6-17 years old group A; 6-35 months old group A; 6-35 months old group D
Biological: high-dose Norovirus Bivalent (GI.1 / GII.4) Vaccine — Intramuscular injection of high-dose Norovirus Bivalent (GI.1 / GII.4) Vaccine in the deltoid muscle of the upper arm
  Arms: 18-59 years old group B; 3-5 years old group B; 6-17 years old group B; 6-35 months old group B; 6-35 months old group E
Biological: placebo — Intramuscular injection of placebo in the deltoid muscle of the upper arm
  Arms: 18-59 years old group C; 3-5 years old group C; 6-17 years old group C; 6-35 months old group C; 6-35 months old group F

SUMMARY:
Phase II clinical study will explore dose and safety, immunogenicity in 4 age groups, including 18-59 years old group, 6-17 years old group, 3-5 years old group, 6-35 months old group, with a total of 1716 subjects.

ELIGIBILITY:
Inclusion Criteria:

* Age range: healthy people aged 6 months -59 years and and older who can provide legal identification;
* Inquired about medical history and physical examination, the investigator judged that the health condition is good;
* The subject and/or his legal guardian and/or his entrusted person can understand the study procedures and informed consent, voluntarily sign informed consent form, and be able to comply with the requirements of the clinical study protocol;
* Females of childbearing age (menarche to menopause) are not pregnant at the time of enrollment (negative urine pregnancy test), not breastfeeding, and have no birth plan within 12 months after enrollment; effective contraception will be taken within 2 weeks before enrollment;

Exclusion Criteria:

First Dose Exclusion Criteria：

* Axillary body temperature is not less than 37.3℃ (older than 14 years) before vaccination, and axillary body temperature is not less than 37.5℃ (14 years or younger) before vaccination;
* Congenital malformations or developmental disorders, genetic defects, severe malnutrition, etc;
* Have received immune enhancement or inhibitor therapy within 3 months (continuous oral or instillation for more than 14 days);
* Have been diagnosed with congenital or acquired immunodeficiency, HIV infection, lymphoma, leukemia or other autoimmune diseases;
* Having serious congenital malformations or chronic diseases (including but not limited to:Down syndrome, thalassemia, heart disease, kidney disease, diabetes, autoimmune disease, genetic allergies, Guillain Barre syndrome, etc.);
* Asthenia or splenectomy, functional asthenia caused by any situation;
* Severe liver and kidney disease, severe cardiovascular disease, drug-uncontrollable hypertension (systolic blood pressure is not less than 140mmHg, diastolic blood pressure is not less than 90mmHg), high blood glucose, diabetic complications , Malignant tumors, various acute diseases or acute attacks of chronic diseases;
* Have a history of chronic gastrointestinal disease, current diarrhea or other digestive system diseases, gastroenteritis requiring treatment in the past 7 days;
* Have a history of abnormal coagulation function (such as coagulation factor deficiency, coagulopathy);
* Have a history of severe allergic reactions to vaccination; allergic to any component of the experimental vaccine
* Have received a live attenuated vaccine within 28 days before vaccination, or received other vaccines（Recombinant vaccine, subunit vaccine, inactivated vaccine） within 14 days before vaccination;
* Received within 6 months before vaccination or plan to receive other study drugs in the near future
* Plan to move before the end of the study or leave the local area for a long time during the scheduled study visit; Other conditions considered by the investigator to be inappropriate for participation in the study.

In addition to the general exclusion criteria, specific populations should also follow the following exclusion criteria:

-Children aged 24 months and under are born prematurely (delivered before the 37th week of pregnancy), low-weight (birth weight for girls <2300g, boys <2500g) infants; Children 24 months of age and younger have a history of dystocia, birth asphyxia or other reasons, a history of neurological damage, severe chronic diseases (such as Down syndrome, sickle cell anemia, or neurological disorders).

Subsequent doses of vaccination Exclusion criteria：

* Have a high fever (axillary temperature is not less than 39.0℃) for three days and severe allergic reaction after the previous dose of vaccination;
* Severe adverse reactions that are causally related to the previous dose of vaccination;
* For those newly discovered or newly identified after the previous dose of vaccine that does not meet the first dose selection criteria or meets the first dose exclusion criteria, the investigator will determine whether to continue participating in the study;
* Other exclusion reasons considered by the investigator.

Ages: 6 Months to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1716 (Estimated)
Dates: Start 2021-06-30 (Actual); Primary Completion 2024-02-28 (Estimated); Study Completion 2024-03-30 (Estimated)

PRIMARY OUTCOMES:
the incidence and severity of any adverse reactions/events within 30 minutes after each dose of vaccination | through 30 minutes after each dose
the incidence and severity of adverse reactions/events within 0-7 days after each dose of vaccination | through 7 days after each dose
the incidence and severity of non-collective adverse reactions/events within 30 days after each dose of vaccination | through 30 days after each dose
  If there is still next vaccination ，collect the incidence and severity of non-collective adverse reactions/events within vaccination interval（28 days） after vaccination
the incidence of SAE from the first dose of vaccination to 6 months after the full course of vaccination | up to 6 months after the full course of vaccination
Antibody titer of HBGA-blocking antibody on the 14th day after the full course of vaccination | 14th day after the full course of vaccination
4-fold Seroconversion rate on the 14th day after the full course of vaccination | 14th day after the full course of vaccination
Antibody titer of（NoV GI.1 and GII.4 HBGA-blocking antibody）on the 14th day after the full course of vaccination | 14th day after the full course of vaccination

SECONDARY OUTCOMES:
Geometric mean Titer of（NoV GI.1 and GII.4 HBGA-blocking antibody）on the 14th day after the full course of vaccination | 14th day after the full course of vaccination
Immune response（compared with before vaccination, the antibody increased by 4 times or more） rate of（NoV GI.1 and GII.4 HBGA-blocking antibody）on the 14th day after the full course of vaccination | 14th day after the full course of vaccination
Antibody titer of（NoV GI.1 and GII.4 HBGA-blocking antibody）on 90th,180th,270th,360th,540th,720th day after the full course of vaccination | 90th,180th,270th,360th,540th,720th day after the full course of vaccination
Binding Antibody (IgG) on 90th,180th,270th,360th,540th,720th day after the full course of vaccination | 90th,180th,270th,360th,540th,720th day after the full course of vaccination

CONTACTS AND LOCATIONS:
Locations (1):
- qixian Center for Disease Control and Prevention, Hebi, Henan, China

IPD SHARING:
Plan to Share IPD: No